CLINICAL TRIAL: NCT03539900
Title: Efficacy and Mechanisms of Naltrexone+Bupropion for Binge Eating Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2000021769; R01DK112771 (NIH)
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Results first posted 2023-07-24 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Binge-Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — bupropion hydrochloride, naltrexone hydrochoride drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NB Medication (Experimental): Bupropion Hydrochloride, Naltrexone Hydrochoride Drug Combination
  Interventions: Drug: Bupropion Hydrochloride, Naltrexone Hydrochoride Drug Combination
- Placebo (Placebo Comparator): Placebo will be inactive and taken daily in pill form.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bupropion Hydrochloride, Naltrexone Hydrochoride Drug Combination — NB medication will combine BUPROPION HYDROCHLORIDE (360 mg/day) and NALTREXONE HYDROCHLORIDE (32 mg/day). Taken daily in pill form.
  Other Names: Contrave
  Arms: NB Medication
Other: Placebo — Placebo will be inactive and taken daily in pill form.
  Arms: Placebo

SUMMARY:
This study will test the efficacy of naltrexone HCI and bupropion HCI (NB) versus placebo in patients with binge-eating disorder (BED), with or without obesity.

DETAILED DESCRIPTION:
Binge-eating disorder (BED), the most prevalent formal eating disorder, is associated strongly with obesity and bio-psychosocial impairment. Improved treatments for patients with BED are needed that can produce sustained clinical outcomes. This study aims to test the efficacy of Naltrexone/Bupropion (NB; FDA-approved anti-obesity combination medication) for the treatment of BED in patients with and without obesity. The RCT will provide new findings regarding the efficacy of NB medication for reducing binge-eating episodes among patients with BED, for reducing weight among patients with BED and obesity, and whether patients with and without obesity derive differential benefit from NB.

ELIGIBILITY:
Inclusion Criteria:

* Binge eating disorder (full criteria as described in the American Psychiatric Association Diagnostic and Statistical Manual of Mental Disorders, 5th edition);
* BMI in the obesity (BMI >30 and <50) or non-obesity (BMI >21.5 and <29.9) range;
* Available for the duration of the treatment and follow-up (15 months);
* Read, comprehend, and write English at a sufficient level to complete study-related materials.

Exclusion Criteria:

* Currently taking opioid pain medications or drugs; or positive drug screen for opiates
* Currently taking medications that influence eating/weight;
* History of seizures;
* Current substance use disorder or other severe psychiatric disturbance (e.g., suicidality);
* Past or current anorexia nervosa or bulimia nervosa;
* Pregnant or breastfeeding;
* Medical status judged by study physician as contraindication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2023-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Grilo, PhD, Principal Investigator — Yale University; Sherry McKee, PhD, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- NB Medication: Naltrexone Hydrochoride, Bupropion Hydrochloride Drug Combination (NB Medication)
  Bupropion Hydrochloride, Naltrexone Hydrochoride Drug Combination: NB medication will combine BUPROPION HYDROCHLORIDE (360 mg/day) and NALTREXONE HYDROCHLORIDE (32 mg/day). Taken daily in pill form.
Period: Overall Study
Arm/Group | NB Medication | Placebo
Started | 43 | 46
Completed | 38 | 44
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NB Medication | Placebo | Total
Number analyzed (Participants) | 43 | 46 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (14.0) | 46.0 (13.2) | 45.7 (13.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Men | 11 | 13 | 24
  Women | 30 | 33 | 63
  Another gender | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 40 | 43 | 83
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 10 | 17
  White | 31 | 31 | 62
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 43 | 46 | 89
Sexual Orientation [Count of Participants; unit: Participants]
  Heterosexual | 38 | 42 | 80
  Homosexual | 2 | 1 | 3
  Bisexual | 3 | 3 | 6
Education [Count of Participants; unit: Participants]
  High School | 8 | 8 | 16
  Some College | 14 | 20 | 34
  College | 12 | 4 | 16
  More than College | 9 | 14 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Binge Eating Frequency
Description: Binge eating will be assessed by interview (Eating Disorder Examination) and the primary outcome is frequency of binge episodes in the past month, comparing baseline and post-treatment. Change is defined as the change in frequency from baseline to post-treatment."
Time Frame: Post-treatment (3 months)
Measure: Mean (Standard Deviation); unit: binge-eating episodes per month
Arm/Group | NB Medication | Placebo
Number analyzed (Participants) | 43 | 46
binge-eating episodes per month | 6.4 (10.6) | 5.4 (9.6)
Statistical Analysis 1: Comparison: NB Medication vs Placebo; Test type: Superiority — Analyses used all available data. Analyses to compare treatments were all intent-to-treat; p = .44, Mixed Models Analysis; Analyses were performed for all randomized participants. Models also considered weight status as a moderator or predictor

2. Primary Outcome: Percent BMI Change
Description: BMI was calculated using measured height and weight. We report percent BMI change using the following formula: ([BMI at posttreatment] - [BMI at baseline])/[BMI at baseline]. Negative values indicate loss.
Time Frame: Post-treatment (3 months)
Measure: Mean (Standard Deviation); unit: percent BMI change
Arm/Group | NB Medication | Placebo
Number analyzed (Participants) | 43 | 46
percent BMI change | -8.0 (11.3) | -0.5 (8.9)
Statistical Analysis 1: Comparison: NB Medication vs Placebo; Test type: Superiority — Analyses used all available data. Analyses to compare treatments were all intent-to-treat; p = .04, Mixed Models Analysis; Analyses were performed for all randomized participants. Models also considered weight status as a predictor or moderator

3. Secondary Outcome: Change in Binge Eating Frequency
Description: Binge eating will be assessed by interview (Eating Disorder Examination) and the primary outcome is frequency of binge episodes in the past month, comparing post-treatment and 6 month post-treatment follow up. Change is defined as the change in frequency from post-treatment to 6 months post-treatment.
Time Frame: 6 months post-treatment
Measure: Mean (Standard Deviation); unit: binge-eating episodes per month
Arm/Group | NB Medication | Placebo
Number analyzed (Participants) | 24 | 23
binge-eating episodes per month | 4.67 (6.29) | 6.00 (9.54)
Statistical Analysis 1: Comparison: NB Medication vs Placebo; Test type: Superiority; p = .98, ANOVA; Analyses used all available data without imputation

4. Secondary Outcome: Change in Binge Eating Frequency
Description: Binge eating will be assessed by interview (Eating Disorder Examination) and the primary outcome is frequency of binge episodes in the past month, comparing post-treatment and 12 month post-treatment follow up. Change is defined as the change in frequency from post-treatment to 12 months post-treatment.
Time Frame: 12 months post-treatment
Measure: Mean (Standard Deviation); unit: binge-eating episodes per month
Arm/Group | NB Medication | Placebo
Number analyzed (Participants) | 22 | 24
binge-eating episodes per month | 6.36 (14.87) | 5.33 (6.82)
Statistical Analysis 1: Comparison: NB Medication vs Placebo; Test type: Superiority; p = .44, ANOVA; Analyses used all available data without imputation

5. Secondary Outcome: Body Mass Index
Description: BMI was calculated using measured height and weight. We report percent BMI change using the following formula: ([BMI at 6 month followup] - [BMI at posttreatment])/[BMI at posttreatment]. Negative values indicate loss.
Time Frame: 6 months post-treatment
Measure: Mean (Standard Deviation); unit: percent BMI change
Arm/Group | NB Medication | Placebo
Number analyzed (Participants) | 13 | 13
percent BMI change | 0.04 (10.51) | 0.05 (4.28)
Statistical Analysis 1: Comparison: NB Medication vs Placebo; Test type: Superiority; p = .99, ANOVA; Analyses used all available data without imputation

6. Secondary Outcome: Body Mass Index
Description: BMI was calculated using measured height and weight. We report percent BMI change using the following formula: ([BMI at 12 month followup] - [BMI at posttreatment])/[BMI at posttreatment]. Negative values indicate loss.
Time Frame: 12 months post-treatment
Measure: Mean (Standard Deviation); unit: percent BMI change
Arm/Group | NB Medication | Placebo
Number analyzed (Participants) | 10 | 13
percent BMI change | -0.20 (12.18) | 3.43 (7.86)
Statistical Analysis 1: Comparison: NB Medication vs Placebo; Test type: Superiority; p = .40, ANOVA; Analyses used all available data without imputation

ADVERSE EVENTS:
Time Frame: Month 1
Description: Participants were interviewed by research clinicians. For non-serious adverse events that were listed as >5% on the package insert for "Contrave" (naltrexone HCl/ bupropion HCl), we provide the total participants [all available data] who reported the adverse event at month 1.
Arm/Group | NB Medication | Placebo
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/46
Other Adverse Events (participants affected / at risk) | 26/43 | 26/46
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NB Medication (N=43) | Placebo (N=46)
Anxiety (Psychiatric disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 10 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 5
Dizziness (General disorders) | 7 | 4
Dry Mouth (Gastrointestinal disorders) | 14 | 4
Headache (General disorders) | 2 | 9
Insomnia (General disorders) | 2 | 6
Nausea (Gastrointestinal disorders) | 6 | 4
Vomiting (Gastrointestinal disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/00/NCT03539900/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT03539900/ICF_001.pdf